CLINICAL TRIAL: NCT02974426
Title: Phase III Study to Evaluate the Optimal Timing of Postoperative Radiotherapy for High Risk of Locoregional Recurrence Patients With Completely Resected Stage IIIA(N2) Non-Small Cell Lung Cancer
Brief Title: To Evaluate the Optimal Timing of Postoperative Radiotherapy in Patients With IIIA(N2) Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment was delayed and the number of eligible patients significantly declined with the use of neoadjuvant or adjuvant ICIs and TKIs therapies. Thus, this trial was closed due to insufficient accrual.
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shanghai Pulmonary Hospital, Shanghai, China (Other); Fudan University (Other); Shanghai Zhongshan Hospital (Other); Ruijin Hospital (Other); RenJi Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaolong Fu, Director, Department of Radiation Oncology, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DLY201619
Record Dates: First submitted 2016-11-20; First posted 2016-11-28 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Non-small Cell Lung Cancer Stage IIIA; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (PORT-first strategy) (Experimental): Concurrent chemoradiotherapy + sequential chemotherapy or PORT + sequential chemotherapy: Participants in the Arm I will receive PORT at the first day of therapy. For lung adenocarcinoma, the first day of radiotherapy will be administered concurrently with chemotherapy (two cycles of chemotherapy given during radiotherapy); then continue to give two cycles of sequential chemotherapy. For squamous cell lung carcinoma, PORT will be administered first followed by subsequent four cycles of sequential chemotherapy.
  Interventions: Radiation: PORT-first; Drug: Platinum-based two drug chemotherapy (cisplatin/carboplatin + vinorelbine or cisplatin/carboplatin + pemetrexed regimen)
- Arm II (PORT-last strategy) (Active Comparator): Four cycles of chemotherapy + sequential PORT: Participants in the Arm II will receive four cycles of adjuvant chemotherapy and after that, sequential PORT (50.4 Gy, 1.8 Gy once daily over 5.5 weeks) will be administered.
  Interventions: Radiation: PORT-last; Drug: Platinum-based two drug chemotherapy (cisplatin/carboplatin + vinorelbine or cisplatin/carboplatin + pemetrexed regimen)

INTERVENTIONS:
Radiation: PORT-first — PORT administered at the first day of adjuvant therapy, using 3- dimensional conformal or intensity-modulated radiation, total dose of 50.4 Gy, 1.8 Gy once daily over 5.5 weeks.
  Arms: Arm I (PORT-first strategy)
Radiation: PORT-last — PORT administered sequentially after participants received adjuvant chemotherapy for four cycles, using 3- dimensional conformal or intensity-modulated radiation, total dose of 50.4 Gy, 1.8 Gy once daily over 5.5 weeks.
  Arms: Arm II (PORT-last strategy)
Drug: Platinum-based two drug chemotherapy (cisplatin/carboplatin + vinorelbine or cisplatin/carboplatin + pemetrexed regimen) — Cisplatin/ carboplatin + vinorelbine regimen for squamous cell lung carcinoma Cisplatin/carboplatin + pemetrexed regimen for lung adenocarcinoma

SUMMARY:
Rationale: Completely resected non-small cell lung cancer (NSCLC) patients with histologically confirmed N2 disease are a heterogeneous population. After complete resection and postoperative chemotherapy (POCT), 20%-40% of cases have a risk of locoregional recurrence (LRR). Postoperative radiation therapy (PORT) should be an integral component of the multidisciplinary treatment for patients with stage IIIA(N2) disease. Postoperative Radiotherapy (PORT)-first strategy may have an advantage of the early administration of locoregional therapy to the mediastinum, in which the tumor burden is presumed to be higher than that of systematic micrometastases. It is not yet known for subsets with specific prognostic factors that confer higher LRR risks, what is the optimal timing of PORT and how to integrate with POCT (in a sequential fashion or concurrent fashion) when PORT is considered for patients with completely resected stage IIIA(N2) NSCLC.

Purpose: This randomized phase III trial is studying the optimal timing of PORT to evaluate whether the PORT-first strategy (PORT administered first with concurrent or subsequent POCT) may be more effective than the PORT-last strategy (PORT administered sequentially following POCT) in treating high risk of LRR patients with completely resected pathologic stage IIIA(N2) NSCLC.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Primary

   - Investigate the optimal timing of PORT for completely resected pathologic stage IIIa(N2) NSCLC by comparing the disease-free survival of patients with high risk of LRR treated with PORT-first vs PORT-last strategy.
2. Secondary

   * Determine the overall survival of patients treated with these regimens.
   * Compare the locoregional recurrence-free survival in patients treated with these regimens.
   * Compare the distant metastasis-free survival in patients treated with these regimens.
   * Determine patterns of failure in patients treated with these regimens.
   * Determine the toxicity, in particular cardiac and pulmonary toxicity, of these regimens in these patients.
   * Determine the prediction models for locoregional recurrence and brain metastasis based on the clinical, pathological, radiological, genetic, tumor microenvironmental and immunological data.

OUTLINE: This is a multicenter, randomized study. The clinical risk prediction model for LRR has been established based on our large institutional database. On multivariate analysis, heavy cigarette smoking history, cN2 status, and number of involved lymph nodes>4 were independently significant factors predicting high risk of LRR. The Prognostic Index (PI) equation was built including the three categorical variables and coefficients based on their level of significance: PI＝(0.9×smoking history)＋(0.5×clinical N status)＋(0.8×number of involved lymph nodes). Patients with the PI score≥3.5 were considered as high risk of LRR.

Patients are stratified according to participating center, EGFR mutation status (EGFR 19del or 21L858R mutations vs others), and use of pretreatment positron emission tomography scans (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I (PORT-first strategy): Concurrent chemoradiotherapy + sequential POCT or PORT + sequential POCT Participants in the Arm I will receive PORT at the first day of therapy. For lung adenocarcinoma, the first day of radiotherapy will be administered concurrently with POCT (two cycles of chemotherapy given during radiotherapy); then continue to give two cycles of sequential chemotherapy. For squamous cell lung carcinoma, PORT will be administered first followed by subsequent four cycles of sequential POCT.
* Arm II (PORT-last strategy): Four cycles of POCT + sequential PORT Participants in the Arm II will receive four cycles of adjuvant chemotherapy and after that, sequential adjuvant thoracic conformal radiotherapy (50.4 Gy, 1.8 Gy once daily over 5.5 weeks) will be administered.

PROJECTED ACCRUAL: A total of 1094 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years to 75 years;
* Complete resection through a surgical procedure of lobectomy, sleeve lobectomy or bilobectomy with microscopically tumor-free resection margins and margin-negative resection of all gross disease; Has undergone systematic nodal assessment (lymph node dissection or sampling with a minimum of three N2 stations sampled or completely dissected, one of which must be the subcarinal station);
* Histologically proven lung adenocarcinoma or squamous cell lung carcinoma of stage pT1-3N2M0 (according to the TNM classification in the Union for International Cancer Control (UICC) 7th ed.);
* Determined as the postoperative high risk of locoregional recurrence;
* No documented metastases (M1) and/or invasion (T4) by the pretreatment examination or at the time of surgery;
* No prior neoadjuvant therapy (chemotherapy and/or RT);
* No prior adjuvant therapy (chemotherapy and/or RT);
* No severe perioperative complications and expected postoperative lifespan ≥4 months;
* ECOG Performance Status 0-1;
* Voluntarily participated in this study and signed the informed consent form by himself or his agent. Had good compliance with the study procedures, and can cooperate with the relevant examination, treatment and follow-up;

Exclusion Criteria:

* Histologically confirmed large cell carcinoma, adenosquamous carcinoma, sarcomatoid carcinomas, neuroendocrine tumors (small cell carcinoma, large cell neuroendocrine carcinoma, carcinoid tumors, etc.), salivary-gland type tumors, adenomas, papillomas, or other and unclassified carcinomas;
* Patients undergoing pneumonectomy;
* Diagnosed with other prior or concurrent malignancies (neoplasm) except for basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years;
* Patients with severe postoperative complications; and time to beginning of the adjuvant therapy has been more than 2 months from the date of surgery;
* Patients with any severe or uncontrolled systematic disease including severe cardiovascular, liver, kidney, hematopoietic, metabolic disease, or uncontrolled active infection that would preclude study participation;
* Patients with positive mental disorder that would preclude study participation;
* Contradictory to chest radiotherapy;
* Pregnant or nursing women;
* Concurrent other anti-cancer treatment;
* Prior preoperative Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKIs) treatment or other targeted therapy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-11; Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 4 years

SECONDARY OUTCOMES:
Overall survival (OS) | 4 years
Locoregional recurrence-free survival (LRFS) | 4 years
Distant metastasis-free survival (DMFS) | 4 years
Treatment-related adverse event | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Fu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NSCLC Meta-analyses Collaborative Group; Arriagada R, Auperin A, Burdett S, Higgins JP, Johnson DH, Le Chevalier T, Le Pechoux C, Parmar MK, Pignon JP, Souhami RL, Stephens RJ, Stewart LA, Tierney JF, Tribodet H, van Meerbeeck J. Adjuvant chemotherapy, with or without postoperative radiotherapy, in operable non-small-cell lung cancer: two meta-analyses of individual patient data. Lancet. 2010 Apr 10;375(9722):1267-77. doi: 10.1016/S0140-6736(10)60059-1. Epub 2010 Mar 24. PMID 20338627
- [Background] Burdett S, Rydzewska L, Tierney J, Fisher D, Parmar MK, Arriagada R, Pignon JP, Le Pechoux C; PORT Meta-analysis Trialists Group. Postoperative radiotherapy for non-small cell lung cancer. Cochrane Database Syst Rev. 2016 Oct 11;10(10):CD002142. doi: 10.1002/14651858.CD002142.pub4. PMID 27727451
- [Background] Lally BE, Zelterman D, Colasanto JM, Haffty BG, Detterbeck FC, Wilson LD. Postoperative radiotherapy for stage II or III non-small-cell lung cancer using the surveillance, epidemiology, and end results database. J Clin Oncol. 2006 Jul 1;24(19):2998-3006. doi: 10.1200/JCO.2005.04.6110. Epub 2006 Jun 12. PMID 16769986
- [Background] Douillard JY, Rosell R, De Lena M, Riggi M, Hurteloup P, Mahe MA; Adjuvant Navelbine International Trialist Association. Impact of postoperative radiation therapy on survival in patients with complete resection and stage I, II, or IIIA non-small-cell lung cancer treated with adjuvant chemotherapy: the adjuvant Navelbine International Trialist Association (ANITA) Randomized Trial. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):695-701. doi: 10.1016/j.ijrobp.2008.01.044. Epub 2008 Apr 24. PMID 18439766
- [Background] Robinson CG, Patel AP, Bradley JD, DeWees T, Waqar SN, Morgensztern D, Baggstrom MQ, Govindan R, Bell JM, Guthrie TJ, Colditz GA, Crabtree TD, Kreisel D, Krupnick AS, Patterson GA, Meyers BF, Puri V. Postoperative radiotherapy for pathologic N2 non-small-cell lung cancer treated with adjuvant chemotherapy: a review of the National Cancer Data Base. J Clin Oncol. 2015 Mar 10;33(8):870-6. doi: 10.1200/JCO.2014.58.5380. Epub 2015 Feb 9. PMID 25667283
- [Background] Billiet C, Decaluwe H, Peeters S, Vansteenkiste J, Dooms C, Haustermans K, De Leyn P, De Ruysscher D. Modern post-operative radiotherapy for stage III non-small cell lung cancer may improve local control and survival: a meta-analysis. Radiother Oncol. 2014 Jan;110(1):3-8. doi: 10.1016/j.radonc.2013.08.011. Epub 2013 Oct 4. PMID 24100149
- [Background] Feng W, Fu XL, Cai XW, Yang HJ, Wu KL, Fan M, Xiang JQ, Zhang YW, Chen HQ. Patterns of local-regional failure in completely resected stage IIIA(N2) non-small cell lung cancer cases: implications for postoperative radiation therapy clinical target volume design. Int J Radiat Oncol Biol Phys. 2014 Apr 1;88(5):1100-7. doi: 10.1016/j.ijrobp.2013.12.048. Epub 2014 Feb 11. PMID 24529715
- [Background] Feng W, Zhang Q, Fu XL, Cai XW, Zhu ZF, Yang HJ, Xiang JQ, Zhang YW, Chen HQ. The emerging outcome of postoperative radiotherapy for stage IIIA(N2) non-small cell lung cancer patients: based on the three-dimensional conformal radiotherapy technique and institutional standard clinical target volume. BMC Cancer. 2015 May 2;15:348. doi: 10.1186/s12885-015-1326-6. PMID 25934006